CLINICAL TRIAL: NCT03851250
Title: A First in Human, Double-blind, Placebo-controlled, Multicentre Phase I/II Study to Evaluate the Safety, Tolerability and Immune Modulatory Effects of MRx-4DP0004 in Participants Taking Long-term Control Medication for Their Asthma
Brief Title: A Study of MRx-4DP0004 in Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor insolvency
Sponsor: 4D pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRx-4DP0004-I-001
Record Dates: First submitted 2019-01-22; First posted 2019-02-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: MRx-4DP0004; Asthma; Live Biotherapeutic Product
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MRx-4DP0004 (Experimental): MRx-4DP0004 is a Live Biotherapeutic Product containing 10^9 to 10^10 Colony Forming Units.
  Participants randomised to this arm will take 2 capsules twice daily at approximately 12 hour intervals for 12 weeks.
  Interventions: Drug: MRx-4DP0004
- Placebo (Placebo Comparator): Participants randomised to this arm will take 2 capsules of placebo twice daily at approximately 12 hour intervals for 12 weeks.
  All participants will receive placebo in a single blind manner for two weeks in addition to the 12 weeks of double blind treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MRx-4DP0004 — Participants randomised to receive MRx-4DP0004 will take it in addition to their regular asthma medication.
  Arms: MRx-4DP0004
Drug: Placebo — Participants randomised to receive placebo will take it in addition to their regular asthma medication.
  Arms: Placebo

SUMMARY:
This is a multicentre, phase I/II, double-blind, placebo-controlled study of MRx-4DP0004 in participants taking long-term medication for asthma. Participants will take two capsules of MRx-4DP0004 twice daily in addition to their existing asthma medication for 12 weeks. Safety and tolerability and immune modulatory effects of MRx-4DP0004 will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented history and diagnosis of asthma at least 6 months prior to Visit 1.
* Stable current asthma treatment as per GINA steps 2-4 (ICS with or without LABA) for at least 2 months prior to Visit 1.
* ACQ-6 score >1.5 and <=4
* FEV1 >50% of predicted normal
* Following protocol specified contraception requirements.

Exclusion Criteria:

* Non-compliant with prescribed asthma maintenance treatment.
* At significant risk of exposure to a change in environmental sensitising substances during the study.
* Co-morbidities not optimally controlled for the last 3 months or any co-morbidity that may put the subject at risk or influence the outcome of the study.
* Hepatitis B or C or HIV.
* GI fistula, feeding tubes or inflammatory bowel disease.
* GI disease resulting in inability for oral intake, malabsorption syndrome, surgical procedures affecting absorption, uncontrolled inflammatory bowel disease.
* History of life-threatening asthma.
* Systemic corticosteroids within 6 weeks of first dose.
* Allergy to all of ampicillin, clindamycin and imipenem.
* Probiotic supplements.
* Immunosuppression or immunosuppressant medication.
* Use of ICS and LABA as Maintenance and Reliever Therapy.
* Smokers or nicotine users within 3 months of screening.
* Former smokers >15 pack years.
* Systemic antibiotics within 6 weeks of first dose.
* Clinically significant haematology and serum biochemistry.
* Sensitivity to any constituent of IMP.
* Diastolic blood pressure <45 or >90, systolic blood pressure <95 or >155mmHg, Pulse rate <40 or >100 bpm.
* Clinically significant ECGs or structural cardiac abnormalities.
* Any other condition that may interfere with primary objective.
* Receipt of a positive COVID-19 test result within 4 weeks of first dose of IMP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Number of participants in each treatment arm experiencing adverse events | Baseline to Day 127
  Adverse events will be considered alongside other primary outcome measures for assessment of safety and tolerability.
Number of clinically relevant adverse changes in clinical laboratory tests in each treatment arm | Baseline to Day 127
  Clinically relevant adverse changes clinical laboratory tests will be considered alongside other primary outcome measures for assessment of safety and tolerability. Clinical laboratory tests will include clinical chemistry, haematology and urinalysis.
Number of clinically relevant adverse changes in vital signs in each treatment arm | Baseline to Day 127
  Clinically relevant adverse changes in vital signs will be considered alongside other primary outcome measures for assessment of safety and tolerability. Vital signs assessments will include measurement of systolic blood pressure, diastolic blood pressure, oral body temperature and pulse rate.
Number of clinically relevant adverse changes in 12-lead ECGs in each treatment arm | Baseline to Day 127
  The number of participants experiencing clinically relevant adverse changes in Clinically relevant adverse changes in vital signs will be considered alongside other primary outcome measures for assessment of safety and tolerability. ECG assessments will include measurement of PR, QRS, QT and QTcF.

SECONDARY OUTCOMES:
Difference in the mean change in the Asthma Control Questionnaire (ACQ-6) between treatment arms | Baseline to Day 99
  The ACQ-6 consists of 6 questions relating to control of asthma symptoms answered on a 7 point scale. The overall score is the mean of the 6 questions and is rated from 0 (totally controlled) to 6 (severely uncontrolled).
Difference in the number of subjects achieving good asthma control (as defined by an ACQ-6 score <1.0) between treatment arms. | Baseline to Day 99
  The ACQ-6 consists of 6 questions relating to control of asthma symptoms answered on a 7 point scale. The overall score is the mean of the 6 questions and is rated from 0 (totally controlled) to 6 (severely uncontrolled).
Difference in the number of asthma exacerbations between treatment arms | Baseline to Day 99
  To determine if MRx-4DP0004 can reduce the number of asthma exacerbations, the number of participants experiencing an exacerbation will be assessed.
Difference in the number of hospitalisations due to asthma exacerbation between treatment arms | Baseline to Day 99
  To determine if MRx-4DP0004 can reduce the number of hospitalisations due to exacerbation of asthma symptoms, the number of participants who are hospitalised due to an exacerbation will be assessed.
Difference in the change from baseline in Forced Expiratory Volume in 1 second (FEV1) between treatment arms | Baseline to Day 99
  To assess the response to MRx-4DP0004 in respect of changes to FEV1, the change from baseline in FEV1 will be assessed.
Difference in the change from baseline in Peak Expiratory Flow (PEF) between treatment arms | Baseline to Day 99
  To assess the response to MRx-4DP0004 in respect of changes to PEF, the change from baseline in PEF will be assessed.
Difference in the change from baseline in Forced Vital Capacity (FVC) between treatment arms | Baseline to Day 99
  To assess the response to MRx-4DP0004 in respect of changes to FVC, the change from baseline in FVC will be assessed.
Difference in the change from baseline in blood eosinophils between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on levels of eosinophils in blood, the change from baseline in percentage and absolute eosinophil counts will be assessed.
Difference in the change from baseline in blood neutrophils between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on levels of neutrophils in blood, the change from baseline in percentage and absolute neutrophil counts will be assessed.
Difference in the change from baseline in use of short-acting beta agonists (SABAs) between treatment arms | 7 period prior to baseline to 7 day period prior to Day 99
  To assess the effect of MRx-4DP0004 on the use of SABAs, the change from baseline in SABA use will be assessed.
Difference in the mean change from baseline in the Asthma Quality of Life Questionnaire (standardised version) (AQLQ(S)) between treatment arms | Baseline to Day 99
  The AQLQ(S) consists of 32 questions relating to quality of life in relation to asthma answered on a 7 point scale. The overall score is the mean of the 32 questions and is rated from 7 (not impaired at all) to 1 (severely impaired).

OTHER OUTCOMES:
Difference in the change from baseline in faecal microbiota profile between treatment arms | Baseline to Day 99
  Faecal samples will be analysed using the MicroDx (R) platform.
Difference in the change from baseline in Fraction exhaled nitric oxide (FeNO) between treatment arms | Baseline to Day 99
  Changes in participants FeNO concentrations will be assessed over the course of the study.
Difference in the change from baseline in Immunoglobulin E (IgE) between treatment arms | Baseline to Day 99
  Changes in participants serum IgE levels will be assessed over the course of the study.
Difference in the change from baseline in leukotriene E4 between treatment arms | Baseline to Day 99
  Changes in participants urinary leukotriene E4 levels will be assessed over the course of the study.
Difference in the change from baseline in peripheral blood mononuclear cells (PBMCs) between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on PBMCs, changes from baseline in lymphocytes and monocytes will be assessed through measurement of CD3, CD16+56, CD45, CD4, CD19, CD8, CD14, CD15, CD16 and CD64.
Difference in the change from baseline in serum cytokines between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on serum cytokines, changes from baseline in IL-1a, IL-1b, CXCL1, CXCL2, IL-6, IL-8, IL-17A, IL-5, IL-4, IL-13, CCL11/eotaxin and TSLP will be assessed
Difference in the change from baseline in sputum eosinophils (percentage count) between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on levels of eosinophils in induced sputum, changes form baseline in percentage eosinophil count will be assessed for participants in the UK only.
Difference in the change from baseline in sputum eosinophils (absolute count) between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on levels of eosinophils in induced sputum, changes form baseline in absolute eosinophil count will be assessed for participants in the UK only.
Difference in the change from baseline in sputum neutrophils (percentage count) between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on levels of neutrophils in induced sputum, changes form baseline in percentage neutrophil count will be assessed for participants in the UK only.
Difference in the change from baseline in sputum neutrophils (absolute count) between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on levels of neutrophils in induced sputum, changes form baseline in absolute neutrophil count will be assessed for participants in the UK only.
Difference in the change from baseline in sputum microbiota profile between treatment groups | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on induced sputum microbiota, changes from baseline in sputum microbiota will be assessed. Sputum samples will be analysed using the MicroDx (R) platform.
Difference in the change from baseline in sputum cytokine profile between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on induced sputum cytokines, changes from baseline in sputum cytokines will be assessed
Difference in the change from baseline in urine metabolomics profile between treatment arms | Baseline to Day 99
  To assess the effect of MRx-4DP0004 on urine metabolomics, the change from baseline in urine metabolomics will be assessed. Urine samples will be analysed using the MicroDx (R) platform

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brightling, Professor, Principal Investigator — University of Leicester
Locations (4):
- OHSU Allergy and Clinical Immunology Clinic, Portland, Oregon, United States
- United Kingdom (3):
  - Bradford Teaching Hospital, Bradford, West Yorkshire
  - 4D Site Leicester, Leicester
  - 4D Site Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No